CLINICAL TRIAL: NCT03640897
Title: Evaluation of the Safety and Performance of LiNiDERM® in the Prevention of Infant Diaper Rash: a Randomized Clinical Trial
Brief Title: Evaluation of the Safety and Performance of LiNiDERM® in the Prevention of Infant Diaper Rash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Gilbert (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LiNiRash
Record Dates: First submitted 2018-07-16; First posted 2018-08-21 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Diaper Rash
Keywords: Infant diaper rash; Baby wipes; Oleocalcareous liniment
MeSH Terms: conditions — Diaper Rash | interventions — Water

STUDY DESIGN:
Intervention Model Description: A monocentric, prospective, randomized, comparator controlled, parallel groups study conducted under paediatric control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liniderm (Experimental): Oleocalcareous liniment Liniderm:
  The product will be applied on the diaper area by parents/ caregivers at each diaper change.
  Interventions: Device: Liniderm
- Wipes (Active Comparator): Free-fragrance baby wipes The product will be used on the diaper area by parents/ caregivers at each diaper change.
  Interventions: Other: Wipes
- Water (Active Comparator): Water and cotton pads The product will be used on the diaper area by parents/ caregivers at each diaper change.
  Interventions: Other: Water

INTERVENTIONS:
Device: Liniderm — Cleaning of the diaper area with Liniderm at each diaper change during 28 days
  Arms: Liniderm
Other: Wipes — Cleaning of the diaper area with wipes at each diaper change during 28 days
  Arms: Wipes
Other: Water — Cleaning of the diaper area with water and cotton pads at each diaper change during 28 days
  Arms: Water

SUMMARY:
Result of immaturity of the skin and factors promoting maceration and mechanical interactions, Irritant diaper dermatitis (IDD) can manifest as early as the third week of life. IDD is a form of contact dermatitis and is the most common inflammatory dermatitis of the diaper area infants. This dermatitis is very common amongst first year of life.

The IDD is characterized by erythema on the convex surfaces with the skin folds spared (W-shaped erythema) and it can cause considerable pain and stress for infants and can be troublesome for their caregivers.

The development of IDD is multifactorial. The critical step in the development of IDD is the occlusion of the skin under the diaper. The skin in the diaper area is predisposed to irritation by the presence of urine, stool, friction on the skin and presence of a high skin pH (potential Hydrogen).

At the cellular level, there is a gradual disorganization of the lipid layers and later an attack of keratinocytes. Clinically, maceration is followed by an inflammatory reaction.

Hence, infrequent diaper changes create overhydration and maceration of the stratum corneum, which makes the skin more sensitive to friction; this may interfere with the protective barrier function, allowing for the exposure of the lower layers to irritants (mechanical, chemical and infectious).

The removal of maceration and the reduction of friction are the key to prevention. But it is recommended to respect preventive measures, in order to preserve the normal skin condition over the long term. Special care procedures are required to ensure healthy development and to protect the skin from irritation and inflammation, as well as a sense of well-being. Although use of appropriately formulated cleansers and emollients can help maintain the epidermal skin barrier in the diaper region, good hygiene and adequate protection are necessary to prevent skin barrier breakdown, rash and infection. The prevention of IDD includes frequent diaper changing, parent education and cleaning.

LiNiRASH is a monocentric, prospective, randomized, comparator controlled study conducted under paediatric control. 132 infants will be followed in this study for 4 weeks during which their parents will use a specific cleaning method: water and cotton pads or wipes or liniment. The objective of this study is to compare the performance and safety of this 3 cleaning methods on the prevention of infant diaper rash.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 - 36 months, in good health, born at term or up to 1 month before term,
* A skin phototype I- III according to Fitzpatrick scale,
* Wearing diapers daily with at least 2 changes per day and a night port,
* For whom parents have given their written informed consent regarding its participation in this clinical investigation.

Exclusion Criteria:

* Wearing washable or pull-on diapers,
* Presenting a diaper rash (in progress),
* Presenting a cutaneous pathology known,
* Treated actually by phototherapy,
* Presenting a cow's milk protein allergy,
* Under medical treatment which may interfere with studied products and/ or skin in the 4-weeks prior to enrolment.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Number of infants who had at least one episode of diaper rash | 28 days
  Every day, in a daily log, parents/ caregivers will report the presence or not of a diaper rash.
  At the end of the follow-up, the investigator must identify infant who have had at least one episode of diaper rash.

SECONDARY OUTCOMES:
Severity of diaper rash episodes: rating | Continuously for 28 days
  Every day, parents/ caregivers will report the rating of erythema if applicable using an illustrated scale ( 4 points scale).
  The rating scale is: 0 (Normal skin), 1 (Mild erythema/ pink skin), 2 (Severe erythema/ red skin) and 3 (Erythema with skin erosion).
Severity of diaper rash episodes: extent | Continuously for 28 days
  Every day, parents/ caregivers will report the extent of erythema if applicable using an illustrated scale ( 4 points scale).
  The extent scale is: 0 (Healthy skin), 1 (On the folds/ small spread), 2 (On the convexity/ moderate spread) and 3 (Wide spread).
Safety of the cleaning method | Continuously for 28 days
  Every day, parents will report intolerance/ discomfort felt. Also, at each visit, the investigator will carry out a clinical examination of the diaper area; the investigator will assess the tolerance using a 4-points Likert scale.
  The 4-points Likert scale is: Bad (0), Moderate (1), Good (2) or Very good (3)
Skin evaluation on the genital area | 0, 14 and 28 days
  Assessment of the skin integrity using a numeric scale (6 points) by the paediatrician at each visit.
  The numeric scale is: 0 (No rash), 1 (Mild irritation or rash), 2 (Moderate irritation or rash), 3 (Considerable irritation or rash), 4 (Extreme irritation or rash) and 5 (Extreme erythema involving entire area, oozing papules, pustules erosion).
  Skin colour measurements using a Chroma Meter.
Paediatrician satisfaction | 14 and 28 days
  The paediatrician's satisfaction (regarding performance) will be assessed for each infant using a 4-point Likert scale.
  The 4-point Likert scale is: Bad (0), Moderate (1), Good (2) or Very good (3)
Well-being | 0, 14 and 28 days
  The well-being of infant will be assessed by parents at each visit. Questions will be about crying, agitation, tension and scratching (Yes/ No).
Parents satisfaction | 14 and 28 days
  The parents' satisfaction (regarding performance and safety) will be assessed using a 4-point Likert scale.
  The 4-point Likert scale is: Bad (0), Moderate (1), Good (2) or Very good (3)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No